CLINICAL TRIAL: NCT04916652
Title: A First-ever Research Collaboration to Characterize MRI Measured Neural Flexibility Development in Chinese Toddlers
Status: Recruiting | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 20.02.INF
Record Dates: First submitted 2020-10-29; First posted 2021-06-07 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Growth & Development; Brain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- S-26 GOLD/ULTIMA GUM-fed group:: Parent(s) to continue feeding their child S-26 GOLD or ULTIMA GUM during the course of the study.
  We will collect information from parents on the S-26 GOLD/ ULTIMA GUM for a maximum of 2 months prior to the study start and during the course of the study.
  Interventions: Radiation: MRI
- Cow's milk-fed group:: Parent(s) to continue feeding their child cow's milk during the course of the study.
  We will collect information from parents on the cow's milk consumed for a maximum of 2 months prior to the study start and during the course of the study.
  Interventions: Radiation: MRI

INTERVENTIONS:
Radiation: MRI — MRI is a safe, non-invasive, cutting edge imaging technology widely used to study the human brain both internationally (NIH connectome project) and in China (China Brain Project). The Baby Connectome Project (BCP) led by NIH scientists has begun data collection on the structural and functional brain development among American infants (Howell, Styner et al. 2019).

SUMMARY:
The overall objective is to characterize the developmental characteristics of MRI measured neural flexibility, as an index of cognitive flexibility, in Chinese toddlers (32 to 42 months old).

DETAILED DESCRIPTION:
The primary objective of this clinical study is to characterize in Chinese toddlers ages 32 - 42 months old the developmental characteristics of MRI measured neural flexibility, as an index of cognitive flexibility, and to assess a range of executive functions (inhibit, shift, emotional control, working memory, plan/organize) using the Global Executive Composite summary score obtained from the BRIEF-P standardized rating scale.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent has been obtained from the parent/legally acceptable representative.
2. Full-term birth (≥ 37 weeks and ≥ 2.5kg)
3. Typically developing Children aged between 32-34 months (2 years 8 months to 2 years10 month of age) at enrolment
4. Neurotypical development as assessed by interview
5. No major risk factors for learning, neurologic, or psychiatric disorder as assessed by interview [defined as a diagnosed learning neurologic or psychiatric disorder in a first degree relative (e.g. parents, siblings)].
6. Dietary requirement detailed below:

S-26 GOLD or ULTIMA GUM--fed group:

I. Daily consumption of S-26 GOLD or ULTIMA GUM for the last 60 days (2 months) II. Desire of the parent to continue feeding GUM during the course of the study

Cow's milk-fed group:

I. Daily consumption of cow's milk or for the last 60 days (2 months) II. Desire of the parent to continue feeding cow's milk during the course of the study

Exclusion Criteria:

1. Delayed birth ( > 41 weeks gestation) as reported in medical record
2. Birth Weight < 2500 g or small for gestational age (birth weight below the 10th percentile) or large for gestational age (birth weight above the 90th percentile) as reported in medical record
3. History of neurological (e.g., head injury, epilepsy), psychiatric or developmental disorder in the toddler as assessed by interview
4. History of diagnosed neurological (e.g., head injury, epilepsy), psychiatric or developmental disorder in parents or siblings, as assessed by interview
5. In utero exposure to alcohol abuse or illicit substances as defined as diagnosis of current substance use disorder in the biological mother and guidelines set by the American College of Obstetricians and Gynecologists and the Royal College of Physicians
6. Multiple birth as reported in medical record
7. Complicated pregnancy (e.g., preeclampsia, gestational diabetes) as assessed by medical interview/ medical record
8. Abnormal screening laboratory values and studies considered to be clinically significant in the opinion of the Investigator (e.g., metabolic disease screening, neonatal bilirubin)

Ages: 32 Months to 34 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy normal developing Chinese toddlers; minimum number of subjects with successful MRI scans at enrolment and age 42 months: N=60 (≈ 30 fed on S-26 GOLD/ ULTIMA growing-up milk (GUM) and ≈30 fed on cows' milk) with key inclusion as daily consumption of the S-26 GUM or cow's milk for the last 60 days (2 mo).
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-04-06 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Neural flexibility | at baseline and 42 months after baseline
  MRI-derived neural flexibility associated with cognitive flexibility (including anterior cingulate cortex, dorsolateral prefrontal cortex, ventrolateral prefrontal cortex, anterior insula, interior frontal junction, superior parietal lobule, precuneus, intraparietal sulcus, and temporoparietal junction)
Global Executive Composite (GEC) score | at baseline and 42 months of age
  executive functions (inhibit, shift, emotional control, working memory, plan/organize) using the Global Executive Composite summary score obtained from the BRIEF-P standardized rating scale

SECONDARY OUTCOMES:
Brain structure (brain regions volume) | at baseline and 42 months of age
  Brain structure (brain regions volume) measured using MRI, including the hippocampal
Brain structure (cortical surface area) | at baseline and 42 months of age
  Brain structure (cortical surface area) measured using MRI
Brain structure (cortical thickness) | at baseline and 42 months of age
  Brain structure (cortical thickness) measured using MRI
Brain structure (myelination) | at baseline and 42 months of age
  Brain structure (myelination) measured using MRI
Brain function (network topologies) | at baseline and 42 months of age
  Brain functional network topologies of the nine commonly assessed brain functional networks, including the primary visual, secondary visual, visual association, motosensory, default mode, frontoparietal, medial frontal, subcortical and cerebellum networks using MRI
Brain function (connection strengths) | at baseline and 42 months of age
  Brain functional connection strengths of the nine commonly assessed brain functional networks, including the primary visual, secondary visual, visual association, motosensory, default mode, frontoparietal, medial frontal, subcortical and cerebellum networks using MRI
Cognitive flexibility | at baseline and 42 months of age
  Using the Behavior Rating Inventory of Executive Function-Preschool Version (BRIEF-P) parent-completed questionnaire
Children development | at baseline and 42 months of age
  Verbal Comprehension, Visual Spatial, Working Memory, and IQ using Wechsler Preschool and Primary Scale of Intelligence (WPPSI-IV)
School readiness | at 42 months of age
  Using Early Human Capability Index (eHCI)
Children behavior (for toddlers) | at baseline and 42 months of age
  Using the Early Childhood Behavioral Questionnaire (ECBQ)
Curiosity | at baseline and 42 months of age
  Using the Curiosity Questionnaire
Sleep quality | at baseline and 42 months of age
  Sleep quality, duration and efficiency (total sleep time / duration of sleep episode *100) computed using the Brief Infant Sleep Questionnaire (BISQ). In addition, an actigraphy in combination with a sleep diary will be used during home period and their relationship will indicate the sleep quality
Home environment | at baseline and 8 months after baseline
  Using validated Child Feeding Practice Questionnaire. In addition, to complete the feeding and adverse events calendar monthly during home period
Feeding practice | at baseline and 42 months of age
  Using the Early Feeding Practice Questionnaire. In addition, the feeding and adverse events calendar monthly during home period
Fecal microbiota composition | at baseline and 42 months of age
  Measured via the shotgun metagenomics sequencing for species composition and functional pathways through stool samples collected
Cognitive flexibility | at baseline and 42 months of age
  Using the Dimensional Change Card Sort (DCCS) task

OTHER OUTCOMES:
Gastrointestinal tolerance (for toddlers) | at baseline and 42 months of age
  using the Toddler Gut Comfort Questionnaire (TGCQ)
Anthropometry (weight in grams) | at baseline and 42 months of age
  Weight in grams and corresponding weight-for-age Z-score according to the WHO growth standards
Anthropometry (body length in centimeters) | at baseline and 42 months of age
  Length in centimeters and corresponding length-for-age Z-score according to the WHO growth standards
Anthropometry (weight-for-length) | at baseline and 42 months of age
  Corresponding weight-for-length Z-score according to the WHO growth standards
Anthropometry (head circumference in centimeters) | at baseline and 42 months of age
  Head circumference in centimeters and corresponding head-circumference-for-age Z-score according to the WHO growth standards
Anthropometry (BMI) | at baseline and 42 months of age
  Weight and height will be combined to report the BMI (kg/m2) and corresponding BMI-for-age Z-score according to the WHO growth standards
Adverse Events (e.g., type, incidence, severity, seriousness) | from enrollment until 42.5 months of age
  standard AE reporting procedure

CONTACTS AND LOCATIONS:
Overall Officials: Fan Jiang, Principal Investigator — Shanghai Children's Medical Center
Locations (1):
- Shanghai Children's Medical Center, Shanghai, Shanghai Municipality, China